CLINICAL TRIAL: NCT01767922
Title: Multicentre, Double-blind Study Versus Placebo on the Impact and Safety of the Daily Administration of Extramel® 140 IU for 12 Weeks on Perceived Stress, Physical and Intellectual Fatigue, Pain Perception, if Present, and the Impact on the Quality of Life of 70 Subjects Included, of Which 60 That Can be Evaluated
Brief Title: Multicentre, Double-blind Study Versus Placebo on Impact and Safety of Extramel® 140 IU on Perceived Stress, Physical and Intellectual Fatigue, Pain Perception if Present, and the Impact on the Quality of Life
Acronym: Ex Stress II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionov (Industry)
Collaborators: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SE-ISO-2007-01
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Life Stress; Fatigue; Pain; Quality of Life
Keywords: Super-Oxyd-Dismutase; SOD; melon juce; perceived stress
MeSH Terms: conditions — Stress, Psychological; Fatigue; Pain | interventions — Extramel; Superoxide Dismutase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extramel 10 mg - 140 UI SOD (Experimental): This arm receives daily one capsule Extramel 10 mg containing 140 UI of SOD.
  Interventions: Dietary Supplement: Extramel 10 mg - 140 UI SOD
- Placebo - exipients only (Placebo Comparator): This arm receives daily one capsule Placebo containing excipients only.
  Interventions: Dietary Supplement: Placebo - Excipient only

INTERVENTIONS:
Dietary Supplement: Extramel 10 mg - 140 UI SOD — Subjects took one capsule of Extramel® 140 IU, or its corresponding placebo, daily over 12 weeks.
  Each volunteer was seen for the 3 visits:
  * visit V1, so-called inclusion visit (D0),
  * visit V2 at 28 days, tolerance of +/- 3 days, (D28) and
  * visit V3 at 84 days, tolerance of +/- 3 days, (D84).
  Arms: Extramel 10 mg - 140 UI SOD
Dietary Supplement: Placebo - Excipient only
  Arms: Placebo - exipients only

SUMMARY:
Objectives of this Multicentre, double-blind study versus placebo were to evaluate impact and safety of the daily administration of Extramel® 140 IU SOD for 12 weeks on perceived stress, physical and intellectual fatigue, pain perception, if present, and the impact on the quality of life of 70 subjects included with 60 that can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female person using an effective contraceptive method, with a negative urine pregnancy test on the inclusion visit for the women of reproductive age.
* Older than 30 years and younger than 65 years
* BMI ≤ 30
* Score greater than 30 on the Cohen perceived stress scale PSS 14.
* Score between 5 and 20 in the Hamilton anxiety scale (excluding the limits).
* Presenting an impact of stress on at least one of the following domains.

  * pain domain with a score greater than 20 millimeters measured on the visual pain evaluation scale,
  * physical condition domain with a score greater than 50 on the Prevost subjective fatigue scale,
  * the psychical condition domain with a global score below 160 in the Stroop test and the reverse Stroop test.
* Stable professional activity since at least 1 year.
* Completely healthy on the day of inclusion, and not taking any medicinal product or dietary supplement with an anti-stress or anti-pain objective.
* Not taking any herbal tea or drink with an anti-stress or anti-pain objective.
* Accepting not to modify his/her dietary habits.
* Having given his/her free, informed and express consent.
* Capable of understanding the nature of the objectives, the consequences of the study and accepting to comply with the protocol requirements.
* Affiliated with a social security insurance or beneficiary of such an insurance system.

Exclusion Criteria:

* Subject presenting an acute pain or pain considered to be incapacitating by the patient him/herself or the observer physician.
* Subject currently under a chronic or acute treatment indicated for stress or anxiety, irrespective of the treatment.
* Subject currently under a chronic or acute treatment indicated for pain problems, irrespective of the treatment.
* Pregnant and/or breast-feeding women.
* Any person who does not satisfy by definition the inclusion criteria.
* Adult protected by the law.
* Any history of psychiatric disease.
* Any pathology in progress or active in the previous month.
* Any administration of a dietary supplement in progress or in the previous month.
* Any subject who within the 3 months following inclusion is likely to experience a major modification of his/her life rhythm (For example marriage, birth of a child, scheduled hospitalization, important exam, etc.) this is left to the discretion of the investigator.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Perceived Stress : Change from base line in Cohen PSS 14 scale at V2 and V3 | Evaluation performed at inclusion day (V1), after 4 weeks at D28 (V2) and then at the end of study visit on D84 (V3).
  Evaluation performed by Cohen PSS 14 scale. It should be noted that in order to be included the patient had to present a minimum score of 30 on the Cohen scale.

SECONDARY OUTCOMES:
Evaluation of evolution of Physical fatigue | Evaluation performed at inclusion day (V1), after 4 weeks at D28 (V2) and then at the end of study visit on D84 (V3).
  Evaluation performed by Prevost subjective fatigue scale and Ruffier test.
Evaluation of evolution of Intellectual fatigue | Evaluation performed at inclusion day (V1), after 4 weeks at D28 (V2) and then at the end of study visit on D84 (V3).
  Evaluation performed by Stroop test, Reverse Stroop test and 15-words Rey test.
Evaluation of evolution of pain | Evaluation performed at inclusion day (V1), after 4 weeks at D28 (V2) and then at the end of study visit on D84 (V3).
  Evaluation of subjects' perceived chronic pain (if existing), was performed using a simple visual analog scale (VAS).
Evaluation of evolution of subject Quality of life | Evaluation performed at inclusion day (V1), after 4 weeks at D28 (V2) and then at the end of study visit on D84 (V3).
  Evaluation of subjects' quality of life, was performed by using Quality of Life SF36 scale.
Evaluation of evolution of subject Quality of life | Evaluation performed at inclusion day (V1), after 4 weeks at D28 (V2) and then at the end of study visit on D84 (V3).
  Evaluation of subjects' quality of life, was performed by using Hamilton anxiety scale.
Evaluation of evolution of subject Quality of life | Evaluation performed at inclusion day (V1), after 4 weeks at D28 (V2) and then at the end of study visit on D84 (V3).
  Evaluation of subjects' quality of life, was performed by using Personnal stress profile questionnary.

OTHER OUTCOMES:
Evaluation of safety | Global safty evaluation performed at the end of study.
  Assessment of the safety performed by analysis of adverse events that occurred throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry CANTIN, MD, Principal Investigator; Patrick LEPRINCE, MD, Study Chair; Hubert TAUPE, PharmD, Study Director — ISOCLIN

REFERENCES:
- [Derived] Carillon J, Notin C, Schmitt K, Simoneau G, Lacan D. Dietary supplementation with a superoxide dismutase-melon concentrate reduces stress, physical and mental fatigue in healthy people: a randomised, double-blind, placebo-controlled trial. Nutrients. 2014 Jun 19;6(6):2348-59. doi: 10.3390/nu6062348. PMID 24949549